CLINICAL TRIAL: NCT04470167
Title: A Multi-center, Randomized, Independent Evaluator-blinded, Subject-blinded, Placebo-controlled, Phase 1/2 Clinical Study to Evaluate Safety and Efficacy of TPX-115 in Patients With Partial-Thickness Rotator Cuff Tear
Brief Title: Phase 1/2 Clinical Study of TPX-115 in Patients With Partial-Thickness Rotator Cuff Tear
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tego Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TG-TPX-115-20-01
Record Dates: First submitted 2020-07-03; First posted 2020-07-14 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPX-115 (Experimental): Subjects receive ultrasound-guided intratendinous injection of TPX-115
  Interventions: Biological: TPX-115
- Placebo (Placebo Comparator): Subjects receive ultrasound-guided intratendinous placebo injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TPX-115 — Ultrasound-guided intratendinous injection of allogeneic fibroblasts(TPX-115)
  Arms: TPX-115
Other: Placebo — Ultrasound-guided intratendinous placebo injection
  Arms: Placebo

SUMMARY:
Rotator cuff tear is one of the most common shoulder diseases and conservative treatment is commonly used for tears involving ≤50% of tendon thickness. Since conventional conservative treatments are not fundamental to repair tendon tissue, there is a growing need of new therapy to improve structural outcome. This study assesses the safety and efficacy of allogeneic fibroblasts on partial-thickness rotator cuff tear. The primary outcome is change in American Shoulder and Elbow Surgeons (ASES) score at 24 weeks after TPX-115 injection. Secondary outcomes include changes from baseline in Visual Analogue Score (VAS) pain score, functional evaluations including Range of Motion (ROM), Constant Score (CS), ASES score and Simple Shoulder Test (SST) at 4, 12 and 24 weeks after administration and structural evaluation using MRI at 24 weeks after injection.

ELIGIBILITY:
Inclusion Criteria:

Participants must;

1. Be 19 years of age or older.
2. Have partial-thickness rotator cuff tear, ≤50% of tendon thickness or of Ellman grade I, II assessed by MRI.
3. Have unilateral shoulder pain lasting more than 3 months despite conservative treatment and VAS pain score ≥5 at screening.
4. Understand fully the study and voluntarily sign the informed consent for participation in the study.

Exclusion Criteria:

Participants with any of the following conditions will be excluded unless stated otherwise;

1. Have partial-thickness rotator cuff tear larger than 50% of tendon thickness or of Ellman grade III, or full-thickness rotator cuff tear confirmed by MRI.
2. Have prior medical history of shoulder surgery on the torn rotator cuff or the upper part of shoulder within 6 months prior to screening visit (shoulder trauma, fracture, upper cervical spine surgery, etc.).
3. Have had subacromial or intra-articular injections on the affected shoulder within 3 months prior to screening visit.
4. Have had received systemic steroid or immunosuppressive agents within 4 weeks prior to screening visit.
5. Have been diagnosed with the following diseases.

   * Inflammatory joint diseases
   * Other shoulder diseases which may cause shoulder pain or functional disorder
   * Autoimmune diseases
   * Active hepatitis B or C
   * HIV Ab positive
   * Malignant tumors within the last 5 years
   * Coagulopathy
   * Genetic disorders related to fibroblasts of collagen
   * Other serious diseases deemed to affect the results of the study
6. Have allergies to bovine proteins or gentamicin.
7. Be pregnant, breastfeeding, planning pregnancy or unwilling to use of contraceptive suggested in this study.
8. Have participated in other clinical trials and received investigational agents within 4 weeks of this study
9. Be deemed inadequate for the study by investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Change in shoulder score of American Shoulder and Elbow Surgeons (ASES) | 24 weeks
  ASES shoulder score is derived from the Visual Analogue Scale (VAS) score for pain and activities of daily living score. The total score - maximum of 100 points - is weighted 50% for pain and 50% for function.

SECONDARY OUTCOMES:
Change in shoulder score of American Shoulder and Elbow Surgeons (ASES) | 4, 12 weeks
  ASES shoulder score is derived from the Visual Analogue Scale (VAS) score for pain and the activities of daily living score. The total score - maximum of points - is weighted 50% for pain and 50% for function.
Change in pain score of Visual Analogue Scale (VAS) | 4, 12, 24 weeks
  VAS pain score is measured on a scale of 0 (no pain) to 10 (worst pain imaginable).
Change in Range of Motion (ROM) | 4, 12, 24 weeks
  Measurement of ROM for forward elevation, external rotation at 90º abduction, external rotation at side and internal rotation at back.
Change in Constant score (CS) | 4, 12, 24 weeks
  The CS total score (100) = Pain (15) + Activity of Daily Living (20) + Mobility (40) + Strength(25)
Change in Simple Shoulder Test (SST) Score | 4, 12, 24 weeks
  SST assesses functional disability of the shoulder (function related to pain, function/strength and Range of Motion).
Change in tear size on Magnetic Resonance Image (MRI) | 24 weeks
  Tear size is assessed by an independent evaluator.
Change in tendon thickness on Magnetic Resonance Image (MRI) | 24 weeks
  Tendon thickness is assessed by an independent evaluator.
Change in tear/footprint on MRI | 24 weeks
  Ratio of tear lengths to whole footprint length is measured by an independent evaluator.
Change of tendinosis on MRI | 24 weeks
  Tendinosis is assessed with tendinosis grading system by an independent evaluator. (0: normal, 1: mild, 2: moderate, 3: marked)

CONTACTS AND LOCATIONS:
Overall Officials: Joo Han Oh, Ph.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No